CLINICAL TRIAL: NCT02562144
Title: A Randomized Clinical Trial of Cutaneous Xylocaine Spray to Reduce Intravenous Cannulation Pain in Adults
Brief Title: A Clinical Trial of Cutaneous Xylocaine Spray to Reduce Intravenous Cannulation Pain in Adults
Acronym: Xylocaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, J. Datema, Master of Science, Isala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Isala
Record Dates: First submitted 2015-09-17; First posted 2015-09-29 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xylocaine spray (Experimental)
  Interventions: Drug: Xylocaine spray
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xylocaine spray — Cutaneous xylocaine spray before intravenous cannulation.
  Other Names: Bananenspray; Lidocaine spray
  Arms: Xylocaine spray
Drug: Placebo — Cutaneous placebo before intravenous cannulation.
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
The enrolled subjects will get an intravenous cannulation in both elbows. The subject will get before xylocaine spray is placed, the intervention-arm, one intravenous cannulation in one of the elbows, the other intravenous cannulation is placed in the other arm before placebo spray is placed, the control arm. The pain score during insertion of the cannulation, the incidence of adverse events and the success rate and degree of difficulty to place an intravenous cannulation. The subjects and the one who place the cannulations will be blinded to the treatment.

DETAILED DESCRIPTION:
The enrolled subjects will get an intravenous cannulation in both elbows. The influence of the left or right-handedness is reduced by randomizing the arms of the subjects in the placebo group or xylocaine group. The subject will get before xylocaine spray is placed, the intervention-arm, one intravenous cannulation in one of the elbows, the other intravenous cannulation is placed in the other arm before placebo spray is placed, the control arm. The pain score during insertion of the cannulation, the incidence of adverse events and the success rate and degree of difficulty to place an intravenous cannulation. The subjects and the one who place the cannulations will be blinded to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18 or older)
* Signing of the informed consent paper

Exclusion Criteria:

* Allergy for xylocaine
* Pregnancy or breast-feeding
* Peripheral neuropathy
* Analgesics in the last 24 hours
* Skin conditions (eczema, psoriasis, infection, or abrasions)
* Difficulties in verbal communication
* No intravenous access in both elbows possible (eg status after axillary dissection )

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-07 (Actual)

PRIMARY OUTCOMES:
The pain score of the tested subjects during intravenous cannulation | A few seconds after intravenous cannulation
  Visual Analogue Scale (VAS) (0 = no pain, 10 = severe pain)

SECONDARY OUTCOMES:
Complications or adverse reactions of xylocaine spray or placebo spray | 5 minutes after xylocaine spray or placebo and 15 minutes after cannulation
Influence of xylocaine spray in successfully placing an IV cannulation | Before intravenous cannulation
  Is the cannulation easy or difficult to access on a scale, 0 to 10 (0 = easy, 10 = very difficult, almost impossible).
The degree of difficulty in successfully placing an IV cannulation | A few seconds after intravenous cannulation
  Indicate in a scale from 10 (0 = easy, 10 = very difficult, almost impossible) or the cannulation was easy or difficult to access

CONTACTS AND LOCATIONS:
Overall Officials: Joris Datema, Drs, Principal Investigator — Isala Zwolle

IPD SHARING:
Plan to Share IPD: No